CLINICAL TRIAL: NCT05926518
Title: Evaluation of Anti-Xa Levels With Nadroparin as Thrombosis Prophylaxis in COVID-19 and Non-COVID-19 Patients Admitted at the ICU
Brief Title: Anti-Xa Level With Thromboprophylactic Dosage Nadroparin in Critically Ill COVID-19 and Non-COVID-19 Patients
Acronym: NADRO
Status: Completed | Type: Observational
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2020/1725
Record Dates: First submitted 2023-06-05; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Critical Illness; Therapeutic Drug Monitoring; Venous Thromboembolism
MeSH Terms: conditions — Critical Illness; Venous Thromboembolism | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID-19 ICU patients: Patients were administered as standard care once daily nadroparin 5700 IU sc (below 100 kg) or twice daily nadroparin 5700 IU sc (above 100 kg).
  Interventions: Procedure: blood sampling
- non-COVID-19 ICU patients: Patients were administered as standard care once daily nadroparin 2850 IU sc.
  Interventions: Procedure: blood sampling

INTERVENTIONS:
Procedure: blood sampling — Blood sampling for the determination of anti-Xa peak levels 4 hours after administration of nadroparin sc.

SUMMARY:
Primary objective The objective of this study is to compare anti-Xa levels obtained with a standard high dose thrombosis prophylaxis in COVID-19 intensive care-patients compared with anti-Xa levels obtained with a normal dose thrombosis prophylaxis in non-COVID-19 intensive care patients.

Secondary objectives

1. To determine the incidence of anti Xa levels out of range of the established target anti Xa level in both groups.
2. To determine the influence of relevant co-variates on the anti-Xa level in the COVID-19 and non-COVID-19 group.

ELIGIBILITY:
Inclusion Criteria:

* All COVID-19 patients > 18 years admitted at the ICU using nadroparin in a high thrombosis prophylactic dosage of 1 dd 5700 IU or 2 dd 5700 IU sc
* All medical non-COVID-19 patients admitted at the ICU using nadroparin in a standard prophylactic dosage of 1 dd 2850 IU sc.
* Minimum estimated length of stay on the ICU of 4 days

Exclusion Criteria:

o (History of) Heparin Induced Thrombocytopenia and Thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult ICU patients (COVID-19 and non-COVID-19 patients) using nadroparin with the intention of thrombosis prophylaxis are included. Anti Xa activity is determined once per patient at least 3 days (peak level after 4th administration) after admission at the ICU and on nadroparin treatment. No randomization.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-11-23 (Actual)

PRIMARY OUTCOMES:
Evaluation of anti-Xa peak level | 2 years
  U/ml

SECONDARY OUTCOMES:
Percentage of anti-Xa levels within target range | 2 years
  Amount of levels within target range (in %)
Influence of covariates (nadroparin dosage, gender, age, weight, BMI, COVID-19, APACHE IV, vasopressor use, eGFR, fluid balance, CRP) on anti-Xa level | 2 years
  relevant correlation

CONTACTS AND LOCATIONS:
Locations (1):
- Monique de Maat, Arnhem, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided